CLINICAL TRIAL: NCT02332993
Title: Nutritional Regulation of Wound Inflammation: Part III
Acronym: FPP3
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Osato Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20141371
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Negative Pressure Therapy; Wound; Open Wound; Type II Obese Diabetic; Type II Non-Obese Diabetic
Keywords: FPP (Fermented Papaya Preparation); Negative Pressure Therapy; Wound Vac; Wound; Type II Diabetic
MeSH Terms: conditions — Wounds and Injuries | interventions — fermented papaya preparation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Supplementation Group: 15 Type 2 Diabetics receiving Negative Wound Pressure Therapy will receive the FPP supplementation to take 3 times a day for 12 weeks (3g/dose).
  Interventions: Dietary Supplement: FPP
- Control Group: 15 Type 2 Diabetics receiving Negative Wound Pressure Therapy will receive no supplementation for 12 weeks.

INTERVENTIONS:
Dietary Supplement: FPP — Made from Carica papaya and represents a sweet and granular substance available over the counter. FPP possesses antioxidant properties that can provide benefit against age-related complications..
  Other Names: Fermented Papaya Preparation; Immun'Age; Osato
  Groups: Supplementation Group

SUMMARY:
The purpose of this study is to examine the changes that result in the wound healing of a type II Diabetic using Negative Pressure Therapy after 12 weeks of daily supplementation of ImmunAge (Fermented Papaya Preparation (FPP). ImmunAge (FPP) is a supplement made from Carica papaya Linn and is available over the counter. ImmunAge (FPP) is an investigational drug, which means it has not been approved by the U. S. Food and Drug Administration (FDA). Approximately 30 subjects will participate in this study. 15 subjects will take the supplementation and 15 subjects to take no supplementation as the control. The

DETAILED DESCRIPTION:
There are a total of 3 study visits over the course of the 12 weeks of the study that will include procedures such as collection of their wound dressing, imaging, blood draw, and receiving the supplement (if in supplementation group). These visits will occur at weeks 0 (consent signed and first distribution of supplements), 2, 3, and 12. At the initial visit the following will be recorded: birth year, gender, ethnicity, race, women of child bearing age: current form of birth control, negative or positive urine Hcg, current medications (medication, dose, frequency, diagnosis), allergies, past or present medical problems, height and weight, HbA1c value, wound site, wound etiology, Blood pressure, pulse, and if the subjects will be randomized into either the control or supplementation group. Subjects will return one week later for study visit one where their blood pressure and pulse will be recorded and will also have one of the following tests completed as a screen fail for the study: Transcutaneous Oxygen Measurement, Toe Pressure, or Ankle-Brachial Index Test. If the reading is inadequate then the subject will no longer participate in the study. Their wound vac sponge will be collected and imaging will be obtained. Subjects will return for study visit 2 where they will have their blood pressure and pulse recorded, will have a blood draw, wound vac sponge collected and wound imaging obtained. Subjects will be asked to return after 12 weeks of supplementation and will have their blood pressure and pulse recorded and wound imaging obtained. Subjects will be asked to bring any empty packets of the supplement to each visit for compliance and will be given a new supply of supplements at the initial visit, visit 1 and 2. Note, if a subject is discontinued from the negative pressure therapy within 2 weeks of consent then the subject will be dropped from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 30 - 70 years
* Patient must understand and give written informed consent
* Patient must be a Type II Diabetic
* HbA1c ≤9%
* Receiving Negative Pressure Therapy (NPWT)

One or more of the following:

* Transcutaneous Oxygen Measurement >30 mmHg
* ABI (Ankle-Brachial Index) >0.7 and less 1.3
* Toe Pressures >30 mmHg

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks and benefits of the study, i.e. Informed consent will be excluded.
* Patients who are pregnant (all women of childbearing age will have a urine Hcg test upon enrollment and agree upon one of the following forms of contraception for the duration of the study: Abstinence, Hormonal contraception, spermicidal condoms, or either you or your partner having been surgically sterilized)
* Immuno-compromised patients; receiving radiation therapy, chemo, or have gone through transplantation or other conditions with prolonged steroid use
* Patients with clinical signs of soft tissue infection such as fever, erythema, leukocytosis, purulent drainage.
* Antibiotic use 7 days prior to biopsy and cultures
* Current smoker
* Clinically significant kidney or liver disease (dialysis)
* Severe neurologic dysfunction

Females who are pregnant as well as individuals who are therapeutically immuno-compromised will also be excluded in order to minimize the risk to such individuals (and fetus) and to decrease statistical variability and to minimize potential of confounders.

Ages: 30 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Type 2 Diabetic patients that are recieving negative pressure therapy for a wound.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09-08 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Wound Macrophage ROS production and NADPH oxidase expression | 12 weeks
  determine the effect of Oral supplementation of FPP on wound macrophage ROS (reactive oxygen species rod outer segment) production and NADPH oxidase expression (RAC levels) in adult T2DM patients with wounds receiving negative pressure therapy
Wound Fluid inflammatory cytokine levels | 12 weeks
  Determine the effect of oral supplementation of FPP on wound fluid inflammatory cytokine levels in adult Type 2 Diabetics Mellitus patients with wounds receiving negative pressure therapy

SECONDARY OUTCOMES:
Wound macrophage function | 12 weeks
  Association of changes in wound macrophage function with wound area
Wound Macrophage function | 12 weeks
  Associations of change in wound macrophage function with cost of care
Wound Macrophage function | 12 weeks
  Association of change in wound macrophage function with amputation rate

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, Ph.D, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - University East Hospital, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio

REFERENCES:
- [Background] Babior BM. The enzymatic basis for O-.2 production by human neutrophils. Can J Physiol Pharmacol. 1982 Nov;60(11):1353-8. doi: 10.1139/y82-202. PMID 6295574
- [Result] Wheat LJ. Infection and diabetes mellitus. Diabetes Care. 1980 Jan-Feb;3(1):187-97. doi: 10.2337/diacare.3.1.187. PMID 6996964
- [Result] Carton JA, Maradona JA, Nuno FJ, Fernandez-Alvarez R, Perez-Gonzalez F, Asensi V. Diabetes mellitus and bacteraemia: a comparative study between diabetic and non-diabetic patients. Eur J Med. 1992 Sep;1(5):281-7. PMID 1341610
- [Result] Bagdade JD, Root RK, Bulger RJ. Impaired leukocyte function in patients with poorly controlled diabetes. Diabetes. 1974 Jan;23(1):9-15. doi: 10.2337/diab.23.1.9. No abstract available. PMID 4809622
- [Result] Bagdade JD, Nielson KL, Bulger RJ. Reversible abnormalities in phagocytic function in poorly controlled diabetic patients. Am J Med Sci. 1972 Jun;263(6):451-6. doi: 10.1097/00000441-197206000-00005. No abstract available. PMID 4403194
- [Result] Geerlings SE, Hoepelman AI. Immune dysfunction in patients with diabetes mellitus (DM). FEMS Immunol Med Microbiol. 1999 Dec;26(3-4):259-65. doi: 10.1111/j.1574-695X.1999.tb01397.x. PMID 10575137
- [Result] Babior BM. Oxygen-dependent microbial killing by phagocytes (first of two parts). N Engl J Med. 1978 Mar 23;298(12):659-68. doi: 10.1056/NEJM197803232981205. No abstract available. PMID 24176
- [Result] Dandona P, Thusu K, Cook S, Snyder B, Makowski J, Armstrong D, Nicotera T. Oxidative damage to DNA in diabetes mellitus. Lancet. 1996 Feb 17;347(8999):444-5. doi: 10.1016/s0140-6736(96)90013-6. PMID 8618487
- [Result] Chang FY, Shaio MF. Respiratory burst activity of monocytes from patients with non-insulin-dependent diabetes mellitus. Diabetes Res Clin Pract. 1995 Aug;29(2):121-7. doi: 10.1016/0168-8227(95)01123-4. PMID 8591699
- [Result] Anuar NS, Zahari SS, Taib IA, Rahman MT. Effect of green and ripe Carica papaya epicarp extracts on wound healing and during pregnancy. Food Chem Toxicol. 2008 Jul;46(7):2384-9. doi: 10.1016/j.fct.2008.03.025. Epub 2008 Apr 3. PMID 18468758
- [Result] Nau JY. [The Pope and the enlightenment of fermented papaya]. Rev Med Suisse. 2005 Feb 9;1(6):459. No abstract available. French. PMID 15786653
- [Result] Imao K, Wang H, Komatsu M, Hiramatsu M. Free radical scavenging activity of fermented papaya preparation and its effect on lipid peroxide level and superoxide dismutase activity in iron-induced epileptic foci of rats. Biochem Mol Biol Int. 1998 Jun;45(1):11-23. doi: 10.1080/15216549800202392. PMID 9635126
- [Result] Rimbach G, Park YC, Guo Q, Moini H, Qureshi N, Saliou C, Takayama K, Virgili F, Packer L. Nitric oxide synthesis and TNF-alpha secretion in RAW 264.7 macrophages: mode of action of a fermented papaya preparation. Life Sci. 2000 Jun 30;67(6):679-94. doi: 10.1016/s0024-3205(00)00664-0. PMID 12659174
- [Result] Marotta F, Barreto R, Tajiri H, Bertuccelli J, Safran P, Yoshida C, Fesce E. The aging/precancerous gastric mucosa: a pilot nutraceutical trial. Ann N Y Acad Sci. 2004 Jun;1019:195-9. doi: 10.1196/annals.1297.031. PMID 15247013
- [Result] Aruoma OI, Colognato R, Fontana I, Gartlon J, Migliore L, Koike K, Coecke S, Lamy E, Mersch-Sundermann V, Laurenza I, Benzi L, Yoshino F, Kobayashi K, Lee MC. Molecular effects of fermented papaya preparation on oxidative damage, MAP Kinase activation and modulation of the benzo[a]pyrene mediated genotoxicity. Biofactors. 2006;26(2):147-59. doi: 10.1002/biof.5520260205. PMID 16823100
- [Result] Calzuola I, Gianfranceschi GL, Marsili V. Comparative activity of antioxidants from wheat sprouts, Morinda citrifolia, fermented papaya and white tea. Int J Food Sci Nutr. 2006 May-Jun;57(3-4):168-77. doi: 10.1080/09637480600658328. PMID 17127467
- [Result] Marotta F, Pavasuthipaisit K, Yoshida C, Albergati F, Marandola P. Relationship between aging and susceptibility of erythrocytes to oxidative damage: in view of nutraceutical interventions. Rejuvenation Res. 2006 Summer;9(2):227-30. doi: 10.1089/rej.2006.9.227. PMID 16706649
- [Result] Marotta F, Weksler M, Naito Y, Yoshida C, Yoshioka M, Marandola P. Nutraceutical supplementation: effect of a fermented papaya preparation on redox status and DNA damage in healthy elderly individuals and relationship with GSTM1 genotype: a randomized, placebo-controlled, cross-over study. Ann N Y Acad Sci. 2006 May;1067:400-7. doi: 10.1196/annals.1354.057. PMID 16804018
- [Result] Amer J, Goldfarb A, Rachmilewitz EA, Fibach E. Fermented papaya preparation as redox regulator in blood cells of beta-thalassemic mice and patients. Phytother Res. 2008 Jun;22(6):820-8. doi: 10.1002/ptr.2379. PMID 18384199
- [Result] Dawkins G, Hewitt H, Wint Y, Obiefuna PC, Wint B. Antibacterial effects of Carica papaya fruit on common wound organisms. West Indian Med J. 2003 Dec;52(4):290-2. PMID 15040064
- [Result] Gurung S, Skalko-Basnet N. Wound healing properties of Carica papaya latex: in vivo evaluation in mice burn model. J Ethnopharmacol. 2009 Jan 21;121(2):338-41. doi: 10.1016/j.jep.2008.10.030. Epub 2008 Nov 8. PMID 19041705
- [Result] Mikhal'chik EV, Ivanova AV, Anurov MV, Titkova SM, Pen'kov LY, Kharaeva ZF, Korkina LG. Wound-healing effect of papaya-based preparation in experimental thermal trauma. Bull Exp Biol Med. 2004 Jun;137(6):560-2. doi: 10.1023/b:bebm.0000042711.31775.f7. PMID 15455084
- [Result] Nayak SB, Pinto Pereira L, Maharaj D. Wound healing activity of Carica papaya L. in experimentally induced diabetic rats. Indian J Exp Biol. 2007 Aug;45(8):739-43. PMID 17877152
- [Result] Pieper B, Caliri MH. Nontraditional wound care: A review of the evidence for the use of sugar, papaya/papain, and fatty acids. J Wound Ostomy Continence Nurs. 2003 Jul;30(4):175-83. doi: 10.1067/mjw.2003.131. PMID 12851592
- [Result] Khanna S, Biswas S, Shang Y, Collard E, Azad A, Kauh C, Bhasker V, Gordillo GM, Sen CK, Roy S. Macrophage dysfunction impairs resolution of inflammation in the wounds of diabetic mice. PLoS One. 2010 Mar 4;5(3):e9539. doi: 10.1371/journal.pone.0009539. PMID 20209061
- [Result] Collard E, Roy S. Improved function of diabetic wound-site macrophages and accelerated wound closure in response to oral supplementation of a fermented papaya preparation. Antioxid Redox Signal. 2010 Sep 1;13(5):599-606. doi: 10.1089/ars.2009.3039. PMID 20095880
- [Result] Marotta F, Koike K, Lorenzetti A, Naito Y, Fayet F, Shimizu H, Marandola P. Nutraceutical strategy in aging: targeting heat shock protein and inflammatory profile through understanding interleukin-6 polymorphism. Ann N Y Acad Sci. 2007 Nov;1119:196-202. doi: 10.1196/annals.1404.011. PMID 18056967
- [Result] Thiele JJ, Traber MG, Packer L. Depletion of human stratum corneum vitamin E: an early and sensitive in vivo marker of UV induced photo-oxidation. J Invest Dermatol. 1998 May;110(5):756-61. doi: 10.1046/j.1523-1747.1998.00169.x. PMID 9579541
- [Derived] Das A, Dickerson R, Ghatak PD, Gordillo GM, Chaffee S, Saha A, Khanna S, Roy S. May Dietary Supplementation Augment Respiratory Burst in Wound-Site Inflammatory Cells? Antioxid Redox Signal. 2018 Feb 10;28(5):401-405. doi: 10.1089/ars.2017.7304. Epub 2017 Oct 16. PMID 28810801